CLINICAL TRIAL: NCT02271321
Title: The Effects of White Noise on Agitated Behaviors and Cortisol in Saliva Among the Patients With Dementia
Brief Title: The Effects of White Noise on Agitated Behaviors and Cortisol Level in Saliva Among the Patients With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hui Yeh, RN, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1021001
Record Dates: First submitted 2014-10-15; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Dementia
Keywords: dementia; white noise; agitation; saliva cortisol
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): The control group will receive usual care
- experimental group (Experimental): The experimental group will receive 20 minute white noise of the ocean and the sound of running water at 16:00 to 17:00 for four weeks periods.
  Interventions: Other: White noise

INTERVENTIONS:
Other: White noise — White noise is a simple, convenient, non-invasive and effective intervention. it sounds like the sound of running water, ocean or fan operation sounds. In this study, Subjects will receive 20 minute white noise of the ocean and the sound of running water at 16:00 to 17:00 for four weeks periods.
  Arms: experimental group

SUMMARY:
The purpose of this study will be to examine the effects of white noise on agitation and saliva cortisol in elderly with dementia.

DETAILED DESCRIPTION:
Aging society is a global trend. In general, each additional five years for older than 65 years old, doubling the prevalence of dementia, that means is constantly increasing in dementia patients. Dementia elderly often appear negative emotion, memory disorders, sleep disorder and agitated behavior. With the progression of dementia, many patients present "sundown syndrome", which particularly appear agitation, hallucinations, delusions in the evening or at night and even accompanied by delirium and confusion. When the patient increased nocturnal awakenings, and even lead to roam at night and confusion, resulting in stress for families and carers. Therefore, the purpose of this study will to examine the effects of white noise on agitation and saliva cortisol in elderly with dementia. The sample sizes was calculated (Power: 0.8, α level: 0.05, effect size: 0.5) by G-Power statistical software. The estimated number of samples will be 35 cases for each group and the loss following rate of 20% will be considered and then each group will recruite 42 cases. In total, 84 cases will be recruited to participate the study. Four dementia care centers located in central and southern Taiwan will be selected and were randomly assigned to the experimental group (two centers) and the control group (two centers). The experimental group will receive 20 minute white noise of the ocean and the sound of running water at 16:00 to 17:00 for four weeks periods. The control group will receive usual care. Before the intervention and pretest, participants will be collected three days of saliva cortisol and observed agitation behavior for 10 days. After the four weeks of white noise intervention, post-test questionnaire, agitation behavior and saliva cortisol will be collected. The information collected will be entered into the computer SPSS 20.0 software for statistical analysis. White noise is a simple, convenient, non-invasive and effective intervention that hopes to improve the agitation behavior and saliva cortisol levels and improve quality of care for dementia elderly.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* No hearing disorders
* Able to communicate in Mandarin or Taiwanese
* Able to attend the program and fill out inform consent.

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Improve the agitation behavior | Change from baseline in agitation behavior at 1 months
  Agitation behavior will be assessed by Cohen-Mansfield Agitation Inventory (CMAI) including physically nonaggressive behavior (PNAB), physically aggressive behavior (PAGB), verbally nonaggressive behavior (VNAB) and verbally aggressive behavior (VAGB) at two different times: (1) baseline data :before white noise intervention, (2) outcome data: at four weeks post-test.

SECONDARY OUTCOMES:
Improve the cortisol homeostasis | Change from baseline in saliva cortisol at 1 months
  Cortisol concentrations will be measured at two different times: (1)baseline data: before white noise intervention, (2) outcome data: at four weeks post-test.
Improve quality of care | Change from baseline in quality of care at 1 months
  Quality of care will be assessed by ease-of-care inventory at at two different times: (1) baseline data :before white noise intervention, (2) outcome data: at four weeks post-test.
Basic attribute data | Baseline
  Barthel Index, amount of activity, date in nursing home and medication situation.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Lin, PhD., Principal Investigator — Department of Nursing, Hung Kuang University; Shu-Hui Yeh, PhD., Principal Investigator — Chang Bing Show Chwan Memorial Hospital & Central Taiwan University of Science and Technology; Li-Jane Tsai, M.S., Principal Investigator — Kuang Tien General Hospital; Lu-Jen Tsai, M.S., Principal Investigator — Chang Bing Show Chwan Memorial Hospital
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan